CLINICAL TRIAL: NCT03268590
Title: Hyperoxia: An Unrecognized Mechanism for Inducing "Hypoxia-Like" Symptoms
Brief Title: Neuroimaging During Pure Oxygen Breathing
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Responsible Party: Principal Investigator, Michael J. Decker, Associate Professor, Case Western Reserve University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CON215044; FA8650-12-D6280 TO0052 (Other Grant/Funding Number: KBRWyle (for Wright Patterson Air Force Base))
Record Dates: First submitted 2017-08-25; First posted 2017-08-31 (Actual); Results first posted 2019-11-13 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-10

CONDITIONS: Hyperoxia; Hypoxia, Brain; Neurobehavioral Manifestations
Keywords: Hyperoxia; Hypoxia, Brain
MeSH Terms: conditions — Hyperoxia; Hypoxia, Brain; Neurobehavioral Manifestations | interventions — Oxygen

STUDY DESIGN:
Intervention Model Description: All participants will undergo neuroimaging (MRI) with electroencephalographic (EEG) cortical network mapping and cognitive assessments during room air breathing (placebo). Room air (21% inspired oxygen) will be delivered via non-rebreather face mask. Persons will serve as their own control and will next undergo neuroimaging (MRI) with electroencephalographic (EEG) cortical network mapping and cognitive assessments during pure oxygen breathing. Pure oxygen (100% inspired oxygen) will be delivered via non-rebreather face mask
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- All Study Participants (Experimental): Breathing 21% oxygen via non-rebreather face mask followed by breathing 100% oxygen via non-rebreather face mask
  Interventions: Drug: Oxygen

INTERVENTIONS:
Drug: Oxygen — Persons will undergo MRI, EEG, and complete computerized cognitive testing in baseline room air. Persons will then breathe 100% pure oxygen and undergo MRI, EEG, and complete computerized cognitive testing. Persons will serve as their own controls.

SUMMARY:
The investigators will conduct a non-randomized clinical trial to examine the effect of pure oxygen breathing on the brain. The study will compare cerebral blood flow, cortical electrical activity, and cognitive performance in 32 persons during room air (21% oxygen) breathing and pure oxygen (100% oxygen) breathing. Subjects will be used as their own controls. The investigators aim to:

1. Determine whether breathing 100% oxygen changes blood flow through the brain. The investigators will learn whether brain blood flow is increased, decreased or stays the same.
2. Determine if changes that might occur in brain blood flow are also accompanied by changes in the brain's electrical activity (EEG).
3. Learn whether changes in the speed at which the brain processes information (cognitive function) accompany changes in brain blood flow and electrical activity that may be seen.

DETAILED DESCRIPTION:
The investigators will conduct a crossover design clinical trial to compare the effect of room air breathing (21% inspired oxygen) with pure oxygen breathing (100% inspired oxygen) on brain blood flow and cortical electrical activity. The study involves a one-time data collection taking place at University Hospitals Cleveland Medical Center on the Case Western Reserve University campus in Cleveland, Ohio. The investigators will perform neuroimaging (MRI) with electroencephalographic (EEG) cortical network mapping and cognitive assessments in all participants during room air breathing and again while breathing 100% pure oxygen. Oxygen will be delivered through a non-rebreather mask. Arterial blood partial pressure of oxygen (PaO2) will be measured twice, from arterial blood samples drawn during breathing room air prior to the MRI scan and again after 30 minutes of breathing 100% oxygen immediately following neuroimaging. Thus, the investigators will be able to determine if breathing pure oxygen may temporarily change brain blood flow and breathing, leading to changes in cognitive status such as euphoria or slowed reflexes. Information gained in this study may have direct operational relevance by helping us to understand one potential cause of "Unexplained Physiologic Events" that are reported in some aircraft pilots when flying at high altitude. Information gained could lead to development of new gas mixtures for use by personnel working in low oxygen high altitude environments.

ELIGIBILITY:
Inclusion Criteria:

1. Persons recruited from currently approved Human Subject Panel for high altitude studies at Wright Patterson Air Force Base, Dayton, OH. Volunteers will have documentation of past exposure to hypobaric conditions, either from past high-altitude flight, as hypobaric chamber personnel, or as participants in previous/current high altitude studies. Persons without past exposure to hypobaric conditions were also eligible to participate.
2. Height 152.5-195.5 cm, weight 40-135 kg.

Exclusion Criteria:

1. Persons who have contraindications to MRI such as cardiac pacemakers, intracranial aneurysm clips, metallic implants or external clips within 10 mm of the head; implanted metallic devices such as pumps or previously implanted neurostimulation devices; cochlear implants, defibrillators, pacing wires, body piercings that cannot be removed, metal filings such as shrapnel, tattoos on the head and neck, or medical conditions contraindicated for MRI safety.
2. History of claustrophobia

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2018-05-02 (Actual); Study Completion 2018-05-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Decker, PhD, Principal Investigator — Case Western Reserve University
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States

REFERENCES:
- [Background] Gao Y, Goodnough CL, Erokwu BO, Farr GW, Darrah R, Lu L, Dell KM, Yu X, Flask CA. Arterial spin labeling-fast imaging with steady-state free precession (ASL-FISP): a rapid and quantitative perfusion technique for high-field MRI. NMR Biomed. 2014 Aug;27(8):996-1004. doi: 10.1002/nbm.3143. Epub 2014 Jun 3. PMID 24891124
- [Background] Beall CM, Strohl KP, Blangero J, Williams-Blangero S, Decker MJ, Brittenham GM, Goldstein MC. Quantitative genetic analysis of arterial oxygen saturation in Tibetan highlanders. Hum Biol. 1997 Oct;69(5):597-604. PMID 9299881
- [Background] Beall CM, Strohl KP, Blangero J, Williams-Blangero S, Almasy LA, Decker MJ, Worthman CM, Goldstein MC, Vargas E, Villena M, Soria R, Alarcon AM, Gonzales C. Ventilation and hypoxic ventilatory response of Tibetan and Aymara high altitude natives. Am J Phys Anthropol. 1997 Dec;104(4):427-47. doi: 10.1002/(SICI)1096-8644(199712)104:43.0.CO;2-P. PMID 9453694
- [Background] Ma D, Gulani V, Seiberlich N, Liu K, Sunshine JL, Duerk JL, Griswold MA. Magnetic resonance fingerprinting. Nature. 2013 Mar 14;495(7440):187-92. doi: 10.1038/nature11971. PMID 23486058
- [Background] Baekey DM, Feng P, Decker MJ, Strohl KP. Breathing and sleep: measurement methods, genetic influences, and developmental impacts. ILAR J. 2009;50(3):248-61. doi: 10.1093/ilar.50.3.248. PMID 19506312
- [Background] Decker MJ, Tabassum H, Lin JM, Reeves WC. Electroencephalographic correlates of Chronic Fatigue Syndrome. Behav Brain Funct. 2009 Oct 6;5:43. doi: 10.1186/1744-9081-5-43. PMID 19807920
- [Background] Decker MJ, Eyal S, Shinar Z, Fuxman Y, Cahan C, Reeves WC, Baharav A. Validation of ECG-derived sleep architecture and ventilation in sleep apnea and chronic fatigue syndrome. Sleep Breath. 2010 Sep;14(3):233-9. doi: 10.1007/s11325-009-0305-z. Epub 2009 Oct 9. PMID 19816726

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 41 persons responded to study advertisements and were screened for eligibility between September 2017 and April 2018. 33 were studied.
Groups:
- All Study Participants: Persons will undergo MRI, EEG, and complete computerized cognitive testing in baseline room air. Persons will then breathe 100% pure oxygen and undergo MRI, EEG, and complete computerized cognitive testing. Persons will serve as their own controls.
Period: Overall Study
Arm/Group | All Study Participants
Started | 33
Completed | 32 (One participant did not complete MRI due to a previously undiagnosed subdermal metal shard in scalp.)
Not Completed | 1
Not completed — Previously unknown exclusion criteria | 1

BASELINE CHARACTERISTICS:
Population: 33 participants were studied; each served as their own control and received both 21% oxygen and 100% oxygen
Groups:
- All Study Participants: Breathing 21% and 100% oxygen via non-rebreather face mask
  Oxygen: Persons will undergo MRI, EEG, and complete computerized cognitive testing in baseline room air. Persons will next breathe 100% pure oxygen and undergo MRI, EEG, and complete computerized cognitive testing. Persons will serve as their own controls.
Arm/Group | All Study Participants
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.61 (13.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 30
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 33
BMI [Mean (Standard Deviation); unit: kg/m^2] | 26.68 (4.15)

OUTCOME MEASURES:

1. Primary Outcome: Cerebral Blood Flow
Description: Change in brain blood flow from Baseline Room Air breathing (21% inspired oxygen) to Pure Oxygen breathing (100% inspired oxygen). Measured using Magnetic Resonance Imaging (MRI).
Time Frame: Baseline and at 30 minutes
Population: Participants with usable MRI arterial spin labeling (ASL) data
Measure: Mean (Standard Deviation); unit: ml/min/100g tissue
Groups:
- All Study Participants: All Persons will undergo MRI, EEG, and complete computerized cognitive testing in baseline room air. Persons will next breathe 100% pure oxygen and undergo MRI, EEG, and complete computerized cognitive testing. Persons will serve as their own controls.
Arm/Group | All Study Participants
Number analyzed (Participants) | 30
ml/min/100g tissue
  21% oxygen cerebral perfusion | 48.54 (12.78)
  100% oxygen cerebral perfusion | 36.17 (11.97)
Statistical Analysis 1: Comparison: All Study Participants; Test type: Superiority; p < 0.05, t-test, 2 sided

2. Secondary Outcome: Cortical Network Activity
Description: Change in alpha cortical electrical activity in the temporal brain region from Baseline Room Air breathing (21% inspired oxygen) to Pure Oxygen breathing (100% inspired oxygen). Measured using MRI-compatible 64-electrode high-density electroencephalography (EEG).
Time Frame: Baseline and at 30 minutes
Population: Participants with usable MRI ASL (arterial spin labeling) data
Measure: Mean (Standard Error); unit: microvolt/second
Groups:
- All Study Participants: Persons will undergo MRI, EEG, and complete computerized cognitive testing in baseline room air. Persons will next breathe 100% pure oxygen and undergo MRI, EEG, and complete computerized cognitive testing. Persons will serve as their own controls.
Arm/Group | All Study Participants
Number analyzed (Participants) | 30
microvolt/second
  21% oxygen spectral power temporal alpha activity | 6.15 (0.34)
  100% oxygen spectral power temporal alpha activity | 6.75 (0.45)
Statistical Analysis 1: Comparison: All Study Participants; Test type: Superiority; p < 0.05, t-test, 2 sided

3. Secondary Outcome: Cognitive Performance
Description: Change in cognitive performance from Baseline Room Air breathing (21% inspired oxygen) to Pure Oxygen breathing (100% inspired oxygen). Measured using the General Cognitive Function score on the MicroCog^TM Assessment of Cognitive Functioning (TM= trademark of Pearson Education, Inc., New York, NY). The computer-administered MicroCog measures changes in cognitive performance in 9 domains related to attention, memory, reasoning, spatial processing, and reaction time. The General Cognitive Function score is a summed score and measures accuracy and speed processing. Education-adjusted Standardized Scores used to compare each study participant against population norms. Higher scores are indicative of better performance. Index Standardized Scores of 69 and below are considered Below Average; scores of 70-84 are considered Low Average; scores of 85-114 are considered to be Average; and scores of 115 and above are considered to be Above Average.
Time Frame: Baseline and at 30 minutes
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | All Study Participants
Number analyzed (Participants) | 30
score on a scale
  21% oxygen cognitive assessment | 97.91 (2.22)
  100% oxygen cognitive assessment | 221.70 (2.49)
Statistical Analysis 1: Comparison: All Study Participants; Test type: Superiority; p < 0.05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 7 days
Description: The participants were healthy and received 100% oxygen. Oxygen is routinely used by healthy persons engaged in certain occupations such as firefighters and high altitude aviators and its use is not considered to be a contributor to all-cause mortality.
Groups:
- All Study Participants When Breathing Room Air; All Study Participants When Breathing Pure Oxygen: Persons will undergo MRI, EEG, and complete computerized cognitive testing in baseline room air. Persons will then breathe 100% pure oxygen and undergo MRI, EEG, and complete computerized cognitive testing. Persons will serve as their own controls.
Arm/Group | All Study Participants When Breathing Room Air | All Study Participants When Breathing Pure Oxygen
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 0/33 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Funding source is the United States Air Force Research Laboratories. The AFRL must approve any presentation or publication of the study results before they can be disseminated.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-06): https://cdn.clinicaltrials.gov/large-docs/90/NCT03268590/Prot_SAP_000.pdf